CLINICAL TRIAL: NCT07186998
Title: The Application of the L Test's Validity and Reliability in Single and Dual Task Conditions in Patients With Multiple Sclerosis
Brief Title: Validity and Reliability of the L Test in Single and Dual Task Conditions in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Physiotherapy and Rehabilitation Department, Assistant Professor, Sanko University
Other Study IDs: hakanpolat6
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Walking; Validity During Daily Activities
Keywords: multiple skleroz; yürüme; geçerlilik; güvenirlilik
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Motor problems and cognitive deficits affecting walking and balance are frequently observed in individuals with MS. As a result of problems occurring in the motor and sensory systems, walking becomes less automatic and greater use is made of cognitive capacity. In addition to deficits in the motor system, individuals with MS experience reduced attention capacity and executive function dysfunction. Walking dysfunction is observed in approximately 85% of MS patients from the early stages, and MS patients report that walking dysfunction significantly limits their daily lives. Gait disorders in individuals with MS are generally characterised by reduced walking speed, shortened stride length, increased double support phase, shortened single support period, cadence changes, and progressively shorter walking distance. MS patients may exhibit variability in walking parameters even in the very early stages. This variability provides information about the extent to which they are at risk of balance impairment and falls. Cognitive impairments are among the most common symptoms of MS. Approximately 65% of individuals with MS report cognitive deficits that emerge in the early stages of the disease. In previous years, motor and cognitive impairments were commonly studied independently of each other. Recently, however, there has been a focus on researching the simultaneous performance of motor and cognitive tasks and revealing the interaction between the two. Performing two actions, motor and cognitive, at the same time can lead to a decrease in performance in one or both actions. This decrease in performance is called Cognitive-Motor Matching. It is usually assessed using dual-task activities that involve motor (walking, balance task) and cognitive tasks (counting backwards, word generation), and the dual-task cost (DTC) is calculated by taking the percentage change in dual-task performance compared to single-task performance. As daily living activities do not involve isolated motor or cognitive tasks, it is recommended in clinical practice and research that both tasks be examined together to calculate the dual-task cost. Many studies evaluating dual-task performance in individuals with MS have reported that individuals with high disability levels, in particular, show greater dual-task cost than healthy individuals. This increase in motor and cognitive dual-task cost in individuals with MS has been shown to be associated with an increased risk of falling. Therefore, it has been stated that it should be included in routine clinical assessments and that intervention studies involving dual-task activities are needed. Dual task impairment in MS may be due to impaired attention, fatigue, and reduced memory capacity or general cognitive functions not related to the use of different strategies. Studies investigating the effect of dual tasks on walking in individuals with MS have reported that dual tasks increase step length, sway phase duration, and double support period, while decreasing walking speed. In the literature, dual tasks have been assessed using tests such as walking on a straight path, tandem walking, and backward walking. Gait assessment has generally been evaluated in a straightforward, simple, and easy manner, such as the Timed Up and Go (TUG) test, the 10-metre walk test, and the 6-minute walk test. Based on this information, we aimed to evaluate dual tasks using the L test, which is a more complex and potentially challenging test. The L test is a modification of the Timed Up and Go test that extends the walking distance to 6 to 20 metres and requires participants to make turns both clockwise and counterclockwise. The L test is a modified form of the TUG test. The walking path is L-shaped. The L test is a more comprehensive test than the TUG test because it involves a greater walking distance and turning activity in both directions. This test indirectly assesses dynamic balance during walking and turning activities. The L test evaluates the fundamental components of functional mobility, such as balance, transfer, walking, and turning. Based on this information, we aimed to assess the applicability of the L test in individuals with multiple sclerosis to evaluate both cognitive and more complex motor skills during single and dual tasks.

DETAILED DESCRIPTION:
The study included volunteers diagnosed with MS who applied to the Neurology Outpatient Clinic at SANKO University Sani Konukoğlu Application and Research Hospital. Patients who met the inclusion criteria were assessed by Dr Meltem Uzun and Dr Hakan Polat in the application laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, SANKO University. All information gathering and assessments on the evaluation form prepared by the researchers were conducted face-to-face with the patients.

First, the individuals' demographic information and disease information (how many years ago they were diagnosed with MS, EDSS: MS severity score) were recorded.

The L test, Timed Up and Go test, and Timed 25-Step Walk test, which assess walking and mobility functions, were performed by two separate physiotherapists with at least 5 years of experience in this field.

Before the tests were administered, the individuals were given a practical explanation of how the tests would be conducted.

The L test was administered first.

The individuals were seated and rested before the L test. The time taken to complete the activities during the tests was recorded using a stopwatch.

The individuals were not informed of the times recorded. The assessments were conducted over two days, with two sessions per day, at one-week intervals.

On the first day, the first assessor (Dr Meltem Uzun, physiotherapist) conducted the L test during the first session. She then conducted the L test under dual-task conditions. For the dual task, individuals were asked to subtract either odd or even numbers from 100 during the test. Subsequently, the Timed Up and Go Test and the Timed 25-Step Walk Test were conducted. In the other session, the second evaluator (Dr. Fzt. Hakan Polat) performed the L test. Subsequently, the L test was performed under dual-task conditions. On the second day of the evaluation, this time the second evaluator (Dr. Fzt. Hakan Polat) began by administering the L test. Subsequently, the first evaluator (Dr Meltem Uzun) performed the L test three times again. Each test was repeated twice, and the average of the two recorded times was noted.

The evaluations were conducted at the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Sanko University.

The individuals in this study were assessed in the same environment in both sessions.

This was done to minimise the effect of environmental factors on the patients' performance.

The room temperature was normal room temperature, it was sufficiently lit, and the floor of the room was a hard surface.

The assessments lasted a total of 25-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65
* Volunteers participating in the study
* Individuals with an Expanded Disability Status Scale (EDSS) score ≤ 4.

Exclusion Criteria:

* Pregnant or within the first 3 months postpartum,
* Who have received corticosteroid treatment within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with multiple sclerosis at the SANKO University Sani Konukoğlu Application and Research Hospital Neurology Outpatient Clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
The timed up-and-go test: | 1 years
  This test assesses walking speed and turning ability over a specified distance on a flat surface. At the start of the test, individuals sit on a chair. A distance of 3 metres is marked out in front of them. Upon the "start" command, they stand up from their seat, walk 3 metres, turn around, walk back, and sit down. The time taken from the "start" command until they are fully seated is recorded in seconds. A shorter time indicates good functional mobility.
L test: | 1 years
  This test indirectly assesses walking speed and dynamic balance during walking and turning activities. It is a modified version of the TUG test. The walking path is L-shaped. The L test is more comprehensive than the TUG test as it involves a greater walking distance and turning activities in both directions. The L test assesses the fundamental components of functional mobility, such as balance, transfer, walking, and turning. During the test, the individual stands up from a chair, walks 3 metres, turns right, walks 7 metres, then turns back and walks along the same path to sit down on the chair. The measured distance is recorded in metres.
Timed 25-step walking test | 1 years
  This test is performed to assess mobility and leg function by recording walking speed over a specified straight distance. Individuals are asked to walk 7.62 metres at their maximum speed on a flat surface in a safe manner. If necessary, individuals are permitted to use walking aids. Participants are asked to walk three times. The average of the times is recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko Unıversıty, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed